CLINICAL TRIAL: NCT06812975
Title: Early Identification of Right Ventricular Dysfunction and Failure in Cardiothoracic and Liver Surgical Patients
Brief Title: Paceport Swan-Ganz Data Collection Study
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: ANES-2020-29144
Record Dates: First submitted 2025-02-02; First posted 2025-02-06 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: RV Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: undergoing any cardiac surgery with cardiopulmonary bypass (CPB) or liver transplantation
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study

SUMMARY:
In association with Edwards LifeSciences, the study will aim to develop an algorithm based on right heart (right atrial, right ventricular and pulmonary artery) waveforms for the early detection of RV dysfunction in cardiothoracic and liver surgery patients at UMMC. This is a prospective, non-interventional, observational study.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥ 18 years of age presenting to the University of Minnesota Medical Center undergoing any cardiac surgery with cardiopulmonary bypass (CPB) or liver transplantation
2. Participate in the Informed Consent process and sign/date the approved informed consent forms
3. Projected to receive Swan-Ganz paceport catheter as part of procedure/standard of care with intermittent cardiac output and mixed venous oxygen saturation (SvO2) measures

Exclusion Criteria:

1. Patients with a history of internal jugular vein thrombosis or known reasons for not being able to thread a central venous catheter through either internal jugular vein
2. Patients with a history of known esophageal strictures, esophageal or stomach cancer, esophageal varices, or any patient in whom a TEE is contraindicated
3. Patients with permanent pacemakers whose right ventricle is being paced and not in normal sinus rhythm
4. Patients unable to consent to participating in the study
5. Patients who are pregnant will be excluded, as part of standard care, all female patients are screened for pregnancy prior to surgery
6. Patients under the age of 18 years old
7. Patients with left bundle branch block, recurrent sepsis, or hypercoagulopathy
8. Patients allergic to FORE-SIGHT Elite sensor adhesive
9. Patients with latex allergy due to presence of latex in the Swan-Ganz catheter balloon.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ≥ 18 years of age presenting to the University of Minnesota Medical Center undergoing any cardiac surgery with cardiopulmonary bypass (CPB) or liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2021-09-18 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
Arterial waveform | 24 hours postoperative
  The slope of the diastolic right ventricular waveform which includes measures of RV end-diastolic pressure and RV contractility (dPdt)

CONTACTS AND LOCATIONS:
Overall Officials: Tjorvi E Perry, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States